CLINICAL TRIAL: NCT05708846
Title: Observational Study for the Improvement of a Digital Health Platform for Remote Monitoring of Patients With Heart Failure
Brief Title: Improvement of a Digital Health Platform for Remote Monitoring of Patients With Heart Failure
Acronym: DHEART
Status: Completed | Type: Observational
Sponsor: humanITcare (Network)
Collaborators: European Innovation Council (Other); Hospital Universitario de Torrevieja (Unknown); University of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: FOLLOWHEALTH-2023-01
Record Dates: First submitted 2023-01-13; First posted 2023-02-01 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Telemonitoring; Remote monitoring; Remote care; Healthcare; Home care; Artificial Intelligence; Chronic patients
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Failure patients telemonitored: Patients will be monitored with the vitalera app and platform
  Interventions: Other: Telemonitoring

INTERVENTIONS:
Other: Telemonitoring — All patients will be telemonitored in order to create a labeled and diverse dataset that will include the following data:
  Physiological parameters (measured periodically), socio-demographic data, risk factors, medication tracking, symptomatology questionnaire for patients, NYHA-class, clinical interventions, health questionnaire answers, classified alarms with their respective timestamp and annotation by the MD, and measurement ranges for each personalized alarm and their changes

SUMMARY:
In the present project, we propose to run an observational study in order to create a huge dataset with telemonitoring data from heart failure (HF) patients. The dataset will contain physiological measurements, socio-demographic data, risk factor information, medication tracking, symptomatology, clinical events and health-related questionnaire answers from each patient. Furthermore, health-related alarms will be delivered to the medical professionals whenever a measure from a patient is out of a predefined clinical range. These alarms and its defined level of relevance (indicated by the medical professionals) will also be Included in the dataset. With the annotated dataset we will be able to implement and train Machine Learning (ML) models that will improve the alarm-based system by making it more robust, trustworthy and reliable.

DETAILED DESCRIPTION:
Heart Failure (HF) is a prevalent and fatal clinical syndrome that affects the quality of life of millions of people worldwide. Between 17% and 45% of patients suffering from HF die within the first year and the remaining die within 5 years. Furthermore, those patients have a high risk of rehospitalization, their associated healthcare costs are huge, and the higher the life expectancy, the higher the disease's prevalence. HF symptoms commonly include shortness of breath, excessive tiredness, and leg swelling which may be worsened with decompensation, and thus displacement to medical centers represents a handicap for such individuals. Remote monitoring technologies provide a feasible solution that allows earlier decompensation identification and better adherence to lifestyle changes and medication. Although telemonitoring by smartphones showed the potential to reduce both the frequency and the duration of HF hospitalizations, there was no association with the reduction of all-cause mortality. Thus, it indicates there is a need to look for more effective and precise methodologies. In recent years, the use of wearable devices that allow daily monitoring of patient's physiological data combined with Artificial Intelligence (AI) has shown immense potential in predicting cardiovascular-related diseases, their adverse events and patient's health status, including that of patients with HF.

Vitalera has implemented a cloud platform and an alarm-based system for remote monitoring of patients that delivers health alarms when a patient's biomedical measurement is out of a predefined range. The platform relieves clinicians and caretakers of going through each patient's data to check for anomalies, accelerating the decision-making process and reducing hospital consultations. However, the system is creating many straightforward alarms that are finally being discarded after evaluation by the medical professional. In the present project, we propose to run an observational study in order to create a huge dataset with patients' clinical data that will contain annotations regarding the relevance of each alarm. With the annotated dataset we will be able to implement and train Machine Learning (ML) models that will improve the remote monitoring system and its alarm-based system by making it more robust, trustworthy and reliable.

This study is being conducted in the framework of a European project promoted by the European Innovation Council (EIC). An earlier version of the platform was validated in a study conducted in 2020 at Hospital de Torrevieja focused on HF. The rationale for this study is in line with vitalera's goal of incorporating artificial intelligence tools to optimize the digital platform. While this study is focused on the creation of a diverse and labeled dataset and on the development of artificial intelligence event-prediction algorithms, a forthcoming second study will focus on the validation of the algorithms to assess their clinical effectiveness.

This is an observational study involving a European network of hospitals. The study consists of continuous remote patient monitoring using vitalera's digital platform and the supplied devices (tensiometer, wearable, scale and oximeter). For 6 months, a total of 500 patients suffering from HF will have their physiological constants monitored.

Patients will be included in the study based on the eligibility criteria and must complete the informed consent provided. Each hospital will decide when to include their patients according to their particular clinical practice (either in the process of discharge planning or during the first follow-up visit, i.e.. 1 or 2 weeks after discharge). The recruitment period is defined as 6 months. That means patients will be incorporated into the study from its start until the sixth month. The last subject included in the study will then finish the study after one year from the first day of the study. Medical professionals from each hospital will be in charge of recruiting the participants. The recruitment rate is specific for each hospital, and it may vary depending on the month.

There is no power calculation associated with the study since the main objective of the study is to gather a dataset in order to train ML models. Once the algorithms are developed, model performance in terms of accuracy will be evaluated by means of C statistic, the area under the receiver operating characteristic curve, and creation of a calibration plot. Furthermore, the models will be evaluated in terms of fairness and potential bias using metrics including statistical parity, group fairness, equalized odds and predictive equality.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure (HF) patients with NYHA Functional Class >= II (according to 2021 EU guidelines).
* Patients older than 18 years old.
* Patients who have suffered an acute decompensation of HF (first and recurrent) in the 30 days prior to enrollment in the study.
* NT-pro BNP ≥300 pg/ml at the moment of hospitalization for patients without ongoing atrial fibrillation/flutter. If ongoing atrial fibrillation/flutter, NT-pro BNP must be ≥600 pg/mL
* Patients must have had an echocardiogram during their HF hospitalization or in the previous 12 months.
* Prior to initiating any procedures, the hospital will ensure that the patient obtains an informed consent document, if applicable.
* All patients will be eligible regardless of the level of LVEF: HFrEF, HFmrEF, and HFpEF.

Exclusion Criteria:

* Oncology patients with metastasis or with chemotherapy treatment ongoing
* Patients participating in other studies or trials.
* Patients not willing to participate.
* Patients over 150 kg
* Patients who do not use Catalan, Spanish, English, Portuguese, Italian, Dutch, German, Swedish, Hungarian, Romanian or French.
* Patients without a mobile phone
* Patients without internet connexion
* Patients with moderate or severe cognitive impairment without a competent caregiver
* Patients with serious psychiatric illness
* Patients with planned cardiac surgery
* Patients with planned heart transplantation or LVAD implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure patients will be recruited from a diversity of hospitals mainly from Spain but also from countries in the south of Europe and Eastern Europe.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio César MD Blázquez, Principal Investigator — Hospital Universitario de Torrevieja
Locations (7):
- Romania (3):
  - Hospital of Galati, Galati, Galați County
  - Hospital Floreasca, Bucharest
  - Colentina Hospital, Bucharest
- Spain (4):
  - Hospital Universitario de Torrevieja, Torrevieja, Alicante
  - Hospital de Figueres, Figueres, Girona
  - Hospital General Universitario Nuestra Señora del Prado, Talavera de la Reina, Toledo
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tripoliti EE, Papadopoulos TG, Karanasiou GS, Naka KK, Fotiadis DI. Heart Failure: Diagnosis, Severity Estimation and Prediction of Adverse Events Through Machine Learning Techniques. Comput Struct Biotechnol J. 2016 Nov 17;15:26-47. doi: 10.1016/j.csbj.2016.11.001. eCollection 2017. PMID 27942354
- [Background] Authors/Task Force Members:; McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2022 Jan;24(1):4-131. doi: 10.1002/ejhf.2333. PMID 35083827
- [Background] Schiff GD, Fung S, Speroff T, McNutt RA. Decompensated heart failure: symptoms, patterns of onset, and contributing factors. Am J Med. 2003 Jun 1;114(8):625-30. doi: 10.1016/s0002-9343(03)00132-3. PMID 12798449
- [Background] Brahmbhatt DH, Cowie MR. Remote Management of Heart Failure: An Overview of Telemonitoring Technologies. Card Fail Rev. 2019 May 24;5(2):86-92. doi: 10.15420/cfr.2019.5.3. eCollection 2019 May. PMID 31179018
- [Background] Scherr D, Kastner P, Kollmann A, Hallas A, Auer J, Krappinger H, Schuchlenz H, Stark G, Grander W, Jakl G, Schreier G, Fruhwald FM; MOBITEL Investigators. Effect of home-based telemonitoring using mobile phone technology on the outcome of heart failure patients after an episode of acute decompensation: randomized controlled trial. J Med Internet Res. 2009 Aug 17;11(3):e34. doi: 10.2196/jmir.1252. PMID 19687005
- [Background] Koulaouzidis G, Iakovidis DK, Clark AL. Telemonitoring predicts in advance heart failure admissions. Int J Cardiol. 2016 Aug 1;216:78-84. doi: 10.1016/j.ijcard.2016.04.149. Epub 2016 Apr 21. PMID 27140340
- [Background] Koehler F, Winkler S, Schieber M, Sechtem U, Stangl K, Bohm M, Boll H, Baumann G, Honold M, Koehler K, Gelbrich G, Kirwan BA, Anker SD; Telemedical Interventional Monitoring in Heart Failure Investigators. Impact of remote telemedical management on mortality and hospitalizations in ambulatory patients with chronic heart failure: the telemedical interventional monitoring in heart failure study. Circulation. 2011 May 3;123(17):1873-80. doi: 10.1161/CIRCULATIONAHA.111.018473. Epub 2011 Mar 28. PMID 21444883
- [Background] Lee S, Chu Y, Ryu J, Park YJ, Yang S, Koh SB. Artificial Intelligence for Detection of Cardiovascular-Related Diseases from Wearable Devices: A Systematic Review and Meta-Analysis. Yonsei Med J. 2022 Jan;63(Suppl):S93-S107. doi: 10.3349/ymj.2022.63.S93. PMID 35040610
- [Background] Guidi G, Pollonini L, Dacso CC, Iadanza E. A multi-layer monitoring system for clinical management of Congestive Heart Failure. BMC Med Inform Decis Mak. 2015;15 Suppl 3(Suppl 3):S5. doi: 10.1186/1472-6947-15-S3-S5. Epub 2015 Sep 4. PMID 26391638
- [Background] Muller-Nordhorn J, Roll S, Willich SN. Comparison of the short form (SF)-12 health status instrument with the SF-36 in patients with coronary heart disease. Heart. 2004 May;90(5):523-7. doi: 10.1136/hrt.2003.013995. PMID 15084550
- [Background] Jaarsma T, Arestedt KF, Martensson J, Dracup K, Stromberg A. The European Heart Failure Self-care Behaviour scale revised into a nine-item scale (EHFScB-9): a reliable and valid international instrument. Eur J Heart Fail. 2009 Jan;11(1):99-105. doi: 10.1093/eurjhf/hfn007. PMID 19147463
- [Background] Roque NA, Boot WR. A New Tool for Assessing Mobile Device Proficiency in Older Adults: The Mobile Device Proficiency Questionnaire. J Appl Gerontol. 2018 Feb;37(2):131-156. doi: 10.1177/0733464816642582. Epub 2016 Apr 11. PMID 27255686

RESULTS

PARTICIPANT FLOW:
Groups:
- Telemonitored Heart Failure Patients: All patients in the observational study will be telemonitored following the same protocol.
Period: Overall Study
Arm/Group | Telemonitored Heart Failure Patients
Started | 154
Completed | 129
Not Completed | 25
Not completed — Death | 5
Not completed — Withdrawal by Subject | 20

BASELINE CHARACTERISTICS:
Arm/Group | Telemonitored Heart Failure Patients
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 96
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity:: White | 132
  Ethnicity:: Latino | 2
NYHA class [Count of Participants; unit: Participants] — The NYHA Functional Classification assesses heart failure severity based on physical activity limitations and symptoms like dyspnea, fatigue, and palpitations. It guides treatment decisions and monitors progression:
  Class I: No symptoms with ordinary activity. Class II: Slight limitation; symptoms with ordinary activity. Class III: Marked limitation; symptoms with less than ordinary activity. Class IV: Symptoms at rest or with minimal activity.
  Ref: McDonagh, et al. "2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure(...)" European Heart Journal
  Participants
    II | 94
    III | 36
    IV | 4
Level of Ejection Fraction (LVEF) [Count of Participants; unit: Participants] — Left Ventricular Ejection Fraction (LVEF) measures the percentage of blood the left ventricle pumps with each heartbeat, essential for heart failure (HF) classification:
  HFrEF: LVEF ≤ 40% (reduced) HFmrEF: LVEF 41-49% (mildly reduced) HFpEF: LVEF ≥ 50% (preserved) HFimpEF: Previously ≤ 40%, now > 40% with improvement LVEF guides HF diagnosis, treatment, and prognosis. McDonagh, et al. "2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure (...)" European heart journal 42.36 (2021): 3599-3726.
  Participants
    <40 | 87
    40-50 | 21
    >=50 | 26
Employment status [Count of Participants; unit: Participants]
  Retired | 94
  Paid | 32
  None | 4
  Unemployed | 3
  Voluntary | 1
Education level [Count of Participants; unit: Participants]
  Without education | 20
  Primary | 32
  Secondary | 37
  High | 45
The patient has a caretaker? [Count of Participants; unit: Participants]
  Yes | 61
  No | 73
Number of people living with the patient [Mean (Standard Deviation); unit: people] | 2 (1)
Smoker [Count of Participants; unit: Participants]
  Yes | 27
  No | 59
  Ex-smoker | 48
Alcohol use [Count of Participants; unit: Participants]
  Yes | 21
  Yes, occasionally | 71
  No | 42
Diabetes [Count of Participants; unit: Participants]
  Yes | 41
  No | 93
Hypertension [Count of Participants; unit: Participants]
  Yes | 103
  No | 31
History of heart disease [Count of Participants; unit: Participants]
  Yes | 86
  No | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Included in the Dataset
Description: The dataset will contain the data from HF patients being telemonitored. This outcome shows the number of patients from which data will be used to build a dataset to train ML models for patient health prediction.
Time Frame: 6 months
Population: All enrolled patients, except the withdrawn ones, are included in the dataset to train ML models.
Measure: Count of Participants; unit: Participants
Arm/Group | Telemonitored Heart Failure Patients
Number analyzed (Participants) | 134
Participants | 134

2. Primary Outcome: Implement ML Models to Improve the Current Alarm-based System Using the Dataset Created
Description: The models should:
  Provide a relevance level for each new alarm by reducing the number of irrelevant alarms and thus fostering personalized follow-up.
  Be robust across different new hospitals and reliable and fair across different target populations, considering the diverse sociodemographic data that will be available in the dataset.
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Track All Clinical Interventions and Events to be Included in the Database
Description: With the registered information, develop and implement ML event prediction algorithms that will add new self-generated alarms to the system.
  These alarms should forecast:
  Untracked hospital interventions, such as UCI visits or hospital readmissions. Changes of medication with their particular estimated dose. Clinical events, such as mortality.
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Assess Patient and Medical Professional Satisfaction With the Digital Platform
Description: Assess patient and medical professional satisfaction with the digital platform at the study's end by using the "Post-Study Usability Questionnaire" (PSSUQ).
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Mean SUS Score to Assess the Usability of the Digital Platform App
Description: Assess the usability of the digital platform at the end of the study by means of the "System Usability Scale" (SUS). The SUS is a standardized tool used to evaluate the usability of digital platforms through a 10-item questionnaire. Each item is rated on a 5-point Likert scale, ranging from "Strongly Disagree" (1) to "Strongly Agree" (5). Scale from 0 to 100. The higher the score the better usablity.
Time Frame: 6 months
Population: We show the results of the SUS score for the patients that answered the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telemonitored Heart Failure Patients
Number analyzed (Participants) | 73
score on a scale | 69.83 (17.97)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Telemonitored Heart Failure Patients
All-Cause Mortality (participants affected / at risk) | 5/134
Serious Adverse Events (participants affected / at risk) | 18/134
Other Adverse Events (participants affected / at risk) | 3/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telemonitored Heart Failure Patients (N=134)
Hospitalization Heart Failure (Cardiac disorders) | 10 (14) — Hospital readmission due to Heart Failure decompensation
Hospitalization Cardiovascular (Cardiac disorders) | 5 (6) — Hospital readmission due to cardiovascular reasons not related to Heart Failure
Hospitalization non CV (Cardiac disorders) | 3 (3) — Hospital reamission not related to any Cardiovascular reason
Urgent visit with intravenous decongestive therapy (Cardiac disorders) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telemonitored Heart Failure Patients (N=134)
Visit to medical emergencies (Cardiac disorders) | 3 (3) — Visit to medical emergencies

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT05708846/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT05708846/ICF_001.pdf